CLINICAL TRIAL: NCT06642207
Title: Effect of IL17 Inhibitor in Comparison With Anti-TNF- α on Platelet Count and Its Association With Disease Activity in Patients With Ankylosing Spondylitis
Brief Title: Effect of IL17 Inhibitor in Comparison With Anti-TNF in Patients With Ankylosing Spondylitis
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Manar Gamal Abdelfattah, Effect of IL17 Inhibitor in comparison with Anti-TNF- α on Platelet count and its association with disease activity in patients with Ankylosing Spondylitis, Sohag University
Other Study IDs: soh-med-24-09-08ms
Record Dates: First submitted 2024-10-01; First posted 2024-10-15 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Anti-TNF; IL17 Inhibitor; IL17; Platelet; Piology
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group A
  Interventions: Diagnostic Test: CBC
- group B
  Interventions: Diagnostic Test: CBC

INTERVENTIONS:
Diagnostic Test: CBC — to compare platelet count in Ankylosing Spondylitis patients in treatment with Anti-TNF- α and patients with IL17 Inhibitor

SUMMARY:
Ankylosing spondylitis (AS) is a chronic, inflammatory autoimmune disease characterized by axial bone inflammation. The main clinical manifestations include back pain and progressive spinal rigidity, as well as inflammation of the hips, shoulders, and peripheral joints. Also, extra-articular manifestations, such as psoriasis, uveitis, and inflammatory bowel disease (IBD).

Indicators of inflammation such as erythrocyte sedimentation rate (ESR) and Creactive protein (CRP), which are typically elevated in AS patients, particularly when peripheral joints are involved, these tests ultimately do not reflect the disease process and have limited sensitivity and specificity. Disease activity in AS has been measured by the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), which includes only patient-reported measures. The assessment of Spondyloarthritis International society (ASAS) developed a new AS disease activity score (ASDAS) that combines patient-reported assessments with erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP). Although platelets play important functions in hemostasis and thrombosis, their functions in controlling immunity and inflammation have drawn more attention recently. Platelets are known to have a key role in controlling inflammatory processes in a variety of pathological states. Overactivated platelets can induce inflammation, which in turn can increase the risk of the development of atherosclerosis, thrombosis, and cardiovascular disorders. Inflammatory diseases, including inflammatory bowel disease (IBD), have platelets play a crucial role in their development. The first-line recommended treatment for active AS is NSAIDs.

Tumor necrosis factor (TNF) inhibitors have completely changed the therapy options for patients who have not improved despite receiving standard NSAID treatment. TNF inhibitors can, however, cause tolerability problems in certain patients or inadequate responses in others, and their effectiveness may gradually diminish. Interleukin (IL)-17 inhibitors are among the new therapeutic alternatives that are currently accessible for these individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfill the Assessment in Spondyloarthritis International Society (ASAS) classification criteria for Axial Spondyloarthritis.
* Patients with disease duration more than 6 months.
* Patients who failed conventional treatment and on bDMARDs (IL17 or Anti-TNF-α).
* Age above 16 years old.
* Patient cooperative and can answer questions.
* Patients who are able and willing to give written informed consent.

Exclusion Criteria:

* Other rheumatologic or collagen diseases.
* Age below 16 years and above 60 years.
* Uncooperative patients.
* Patient not able and willing to give written informed consent.
* Patient with other causes of platelet dysfunction, count irregularity.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Patients fulfill the Assessment in Spondyloarthritis International Society (ASAS) classification criteria for Axial Spondyloarthritis. [13]
  2. Patients with disease duration more than 6 months.
  3. Patients who failed conventional treatment and on bDMARDs (IL17 or Anti-TNF-α).
  4. Age above 16 years old.
  5. Patient cooperative and can answer questions.
  6. Patients who are able and willing to give written informed consent
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Effect of IL17 Inhibitor in comparison with Anti-TNFα on Platelet count | 6 months
  Evaluate the effect of IL-17 inhibitor and Anti-TNF-αon platelet count in AS patients.
Platelet count association with disease activity in patients with Ankylosing Spondylitis | 6 months
  Platelet count as indicator of disease activity and follow up of AS patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Braun J, Sieper J. Ankylosing spondylitis. Lancet. 2007 Apr 21;369(9570):1379-1390. doi: 10.1016/S0140-6736(07)60635-7. PMID 17448825
- [Background] Molto A, Nikiphorou E. Comorbidities in Spondyloarthritis. Front Med (Lausanne). 2018 Mar 12;5:62. doi: 10.3389/fmed.2018.00062. eCollection 2018. PMID 29594122
- [Background] Reveille JD. Biomarkers for diagnosis, monitoring of progression, and treatment responses in ankylosing spondylitis and axial spondyloarthritis. Clin Rheumatol. 2015 Jun;34(6):1009-18. doi: 10.1007/s10067-015-2949-3. Epub 2015 May 5. PMID 25939520
- [Background] van der Heijde D, Lie E, Kvien TK, Sieper J, Van den Bosch F, Listing J, Braun J, Landewe R; Assessment of SpondyloArthritis international Society (ASAS). ASDAS, a highly discriminatory ASAS-endorsed disease activity score in patients with ankylosing spondylitis. Ann Rheum Dis. 2009 Dec;68(12):1811-8. doi: 10.1136/ard.2008.100826. Epub 2008 Dec 5. PMID 19060001